CLINICAL TRIAL: NCT07198594
Title: A Study on the Efficacy and Safety of Accelerated Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder and Its Underlying Neurological Mechanisms
Brief Title: Accelerated rTMS Therapeutic Approach for Refractory Obsessive-Compulsive Disorder
Acronym: OCDTMS-IFC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University (Other)
Responsible Party: Principal Investigator, zhaoyijie, Associate Professor, Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDJW-KY-2025-017
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Obsessive Compulsive Disorder (OCD); Obsessive - Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS (Experimental): individualized rTMS targeting IFC, with symptom provocation
  Interventions: Other: rTMS

INTERVENTIONS:
Other: rTMS — individualized rTMS target the IFC with symptom provocation

SUMMARY:
The goal of this clinical trial is to learn if individualized accelerated repetitive transcranial magnetic stimulation (rTMS) targeting the inferior frontal cortex combined with symptom provocation works to treat obsessive-compulsive disorders (OCD) in adults. It will also learn about the safety of rTMS over right IFC. The main questions it aims to answer are:

* Does rTMS using a new individualized IFC target relieve participants' OCD symptoms?
* What medical problems do participants have when taking rTMS?

Participants will:

* Take rTMS six times per day for 5 consecutive days
* Visit the clinic once at baseline, the day and four weeks after treatment for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects with Obsessive Compulsive Disorders (OCD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria
* without associated tics ("Gilles de la Tourette" Syndrome)
* Age 18-60 years, right-handed
* Disease severity: Yale-Brown Obsessive Compulsive Scale score ≥16 for OCD patients
* Medication stable for at least 4 weeks
* Resistant patients to standard treatments: partial but insufficient response (reduction of Y-BOCS score < 35%) or lack of response to previous well conducted treatment including: optimal tolerated dose and adequate duration (> 12 weeks) of at least 2 Serotonin Reuptake Inhibitors (selective serotonin reuptake inhibitors, clomipramine), or 1 Serotonin Reuptake Inhibitors + 1 augmentation strategy (adjunction of an antipsychotic - such as risperidone or olanzapine or aripiprazole - or lithium or buspirone)
* No systematic rTMS therapy in the past six months;
* Signature of informed consent form;
* Normal vision or corrected vision;
* Capacity to complete protocol-specified tests.

Exclusion Criteria:

* Abnormal cognitive status (assessed using MoCA with score <24);
* Other primary diagnosis than OCD (comorbid mild depression is tolerated)
* Comorbid diagnosis of schizophrenia/ psychotic disorder, bipolar disorder, substance abuse or dependance3)
* Significant self-harm intent or severe suicidal tendencies within the past year;
* Irreversible visual or auditory impairment preventing completion of scales or related assessments;
* Presence of metallic implants, such as pacemakers or stents;
* Any current or potential medical, psychological, social, or geographical factors compromising patient safety or study participation;
* Poor compliance;
* Claustrophobia;
* History of epilepsy or familial epilepsy
* Pregnant or lactating women (women of childbearing potential must obtain a negative pregnancy test result prior to study commencement and employ medically approved contraceptive measures);
* Deterioration or failure of vital organ function (cardiac, pulmonary, hepatic, renal, etc.); or unstable vital signs;
* Conditions unsuitable for this stimulation site, such as increased intracranial pressure, elevated intraocular pressure, or glaucoma
* History of or concomitant neurological disorders: cerebrovascular disease, central nervous system infections, Creutzfeldt-Jakob disease, Huntington's disease and Parkinson's disease, Lewy body dementia, traumatic brain injury dementia, other physical/chemical factors (drugs, alcohol, CO, etc.), significant somatic diseases (hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space-occupying lesions (subdural haematoma, brain tumours), endocrine system disorders (thyroid disease, parathyroid disease), and dementia caused by vitamin deficiency or any other cause

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
OCD Symptom Severity Assessed by Y-BOCS | From Baseline to 6 months after treatment
  Change from Baseline to 4 weeks after treatment in OCD Symptom Severity

SECONDARY OUTCOMES:
Safety for rTMS targeting IFC | Adverse Events after treatment
  Number of Participants with Treatment-Related Adverse Events
Depression Severity Assessed by HAMD | From baseline to 4 weeks after treatment
Anxitey Severity Assessed by HAMA | From Baseline to 4 weeks after treatment
Clinical Efficacy Assessed by CGI | From Baseline to 4 weeks after treatment
Uncertainty Assessed by IUI and IUS-12 | From Baseline to 4 weeks after treatment
Self-rated Beck Depression Inventory (BDI) | From Baseline to 4 weeks after treatment
Self-rated State-Trait Anxiety Inventory (STAI) | From Baseline to 4 weeks after treatment
Self-rated Short UPPS-P Impulsive Behaviour Scale | From baseline to 4 weeks after treatment
Neuroimaging by Magnetic resonance imaging | From baseline to 4 weeks after treatment
Cognitive Function Assessent by tasks | From baseline to 4 weeks after treatment
  Including Cantab and coded tasks in Matlab

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong New Area Mental Health Centre, Shanghai, Shanghai Municipality, China

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT07198594/Prot_ICF_000.pdf